CLINICAL TRIAL: NCT03224156
Title: Prediction of Sudden Cardiac Death in Dilated Cardiomyopathy: The PREDICT-DCM Trial.
Brief Title: Prediction of Sudden Cardiac Death in Dilated Cardiomyopathy
Acronym: PREDICT-DCM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Marco Ochs, Dr. med. Marco Ochs, University Hospital Heidelberg
Other Study IDs: S-281/2017
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Cardiomyopathy, Dilated; Sudden Cardiac Death
MeSH Terms: conditions — Cardiomyopathy, Dilated; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dilated Cardiomyopathy
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance Imaging — Patients undergo baseline characterisation including CMR, ECG, blood samples prior to ICD implantation.

SUMMARY:
PREDICT-DCM Trial is a multi-centre, prospective observational trial including patients with DCM undergoing cardiac magnetic resonance imaging (CMR) prior to ICD or event recorder implantation.

DETAILED DESCRIPTION:
Prophylactic ICD implantation was recently found to be non-beneficial over usual clinical care in non-ischemic systolic heart failure (LVEF≤35%) and 60-70% percent of SCD cases even occur in individuals with LEVF>35%. A growing evidence, that emphasizes the urgent need to improve the prediction of sudden cardiac death (SCD) in dilated cardiomyopathy (DCM).

CMR provides unique information on myocardial mechanics, fibrotic burden, inflammation and microvascular dysfunction, thereby allowing to quantify key substrates for myocardial arrhythmogenic potential.

PREDICT-DCM Trial is a multi-centre, prospective observational trial including patients with DCM undergoing cardiac magnetic resonance imaging (CMR) prior to ICD or event recorder implantation.

Acquired candidate predictors are among others:

* Global and regional T1/T2
* T1/T2 inhomogeneity
* Extracellular volume fraction
* Microvascular dysfunction
* LA function and filling fraction
* Global and regional circumferential, radial or longitudinal myocardial strain
* Biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Dilated Cardiomyopathy
* ICD Indication
* age ≥ 18 years
* signed informed consent

Exclusion Criteria:

* severe claustrophobia
* rest dyspnea
* tachycardia or severe arrhythmia
* intolerance to gadolinium-based contrast agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Dilated Cardiomyopathy prior to ICD-implantation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Primary Combined Endpoint | 18 months
  Sudden Cardiac Death OR sustained VT OR non-sustained, long run VT

SECONDARY OUTCOMES:
Mortality | 18 months
  Cardiac Death

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Heidelberg, Krehl Klinik, Department of Cardiology, Heidelberg, Baden-Wurttemberg
  - GRN Hospital Weinheim, Weinheim, Baden-Wurttemberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: University Hospital Heidelberg — https://www.heidelberg-university-hospital.com/